CLINICAL TRIAL: NCT05504889
Title: Cholesterol and CYP3A4/5 Metabolism Across Pregnancy and Postpartum
Acronym: CAMCAP
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Sponsor
Other Study IDs: STU00217170
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related
Keywords: pregnancy; CYP3A; postpartum; hydroxycholesterol ratio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endogenous cholesterol, 4-beta-hydroxycholesterol, estradiol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OPTIMOM residual samples: Residual plasma samples collected in one of our prior studies monthly across pregnancy (OPTIMOM, NICHD 1U54HD085601-01, Clinical Trials.gov ID NCT02519790; K. Wisner, PI) will be evaluated for cholesterol and 4β-hydroxycholesterol.
  These samples were obtained from women who gave their consent for use of their blood samples for future studies. All OPTI-MOM participants have been genotyped for variants in CYP3A5 using commercial allelic discrimination assays (ThermoFisher Scientific, Waltham, MA, with Taqman probes.)
- Newly recruited subjects: Plasma samples will be collected from newly recruited subjects.

SUMMARY:
This study addresses the second aim of the grant (R01 HD0899455), which is to determine temporal changes in CYP3A4-mediated drug metabolism sequentially across pregnancy and after birth.

DETAILED DESCRIPTION:
This study addresses the second aim of the grant (R01 HD0899455), which is to determine temporal changes in CYP3A4-mediated drug metabolism sequentially across pregnancy and after birth.

In studies with human hepatocytes, we found that serum from women in the first trimester led to the highest CYP3A4 expression compared to those from the second or third trimester or after birth. Among the hormones with elevated plasma concentrations in early pregnancy, our studies revealed that thyroid hormone enhances CYP3A4 expression in human hepatocytes. Based on the results, we hypothesized that CYP3A4-mediated drug metabolism is highest during early pregnancy (compared to the later time points of pregnancy or postpartum period) in part due to changes in thyroid hormone concentration.

To test this hypothesis, we will evaluate the conversion of endogenous cholesterol to its 4β-hydroxycholesterol metabolite, which is facilitated by CYP3A4. To assess additional factors that affect CYP3A activity, we will obtain DNA. About 75% of African Americans, but only 10-20% of people of European descent, carry the active allele CYP3A5*1, which significantly increases the clearance of many CYP3A4/5 substrates, including the conversion of cholesterol to 4β-hydroxycholesterol.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Pregnant before 14w0d OR postpartum between before 18w0d
* Singleton gestation (as this will result in more consistent inter-individual measures)

Exclusion Criteria:

* Chronic use of compounds that are substrates or inhibitors of CYP3A4 inhibitors, which will interfere with the concentrations and ratio. Potent inhibitors include clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil, goldenseal and grapefruit. Inducers of CYP3A4 include phenobarbital, phenytoin, rifampicin, St. John's Wort and glucocorticoids.
* Diagnosis of alcoholism or substance use.
* Covid infection or within 4 weeks of positive test due to possible effect on hepatic function

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample of pregnant or postpartum woman in areas surrounding Chicago, IL.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the endogenous metabolic ratio of 4β-hydroxycholesterol to cholesterol (4β-OHC/C, a marker of CYP3A activity) from early pregnancy through 17 weeks 6 days after delivery | Between 4-13 weeks of pregnancy, and 1-18 weeks postpartum
  plasma concentrations

SECONDARY OUTCOMES:
Impact of active CYP3A5 phenotype on the 4β-hydroxycholesterol to cholesterol metabolic ratio | Between 4-13 weeks of pregnancy, and 1-18 weeks postpartum
  plasma concentrations
Impact of estradiol concentrations on ratio in the early first trimester of pregnancy | Between 4-13 weeks of pregnancy, and 1-18 weeks postpartum
  plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Wisner, M.D., M.S., Principal Investigator — Northwestern University; Hyunyoung Jeong, PharmD, PhD, Principal Investigator — Purdue University; Catherine S Stika, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Asher Center for the Study and Treatment of Depressive Disorders, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bjorkhem-Bergman L, Backstrom T, Nylen H, Ronquist-Nii Y, Bredberg E, Andersson TB, Bertilsson L, Diczfalusy U. Comparison of endogenous 4beta-hydroxycholesterol with midazolam as markers for CYP3A4 induction by rifampicin. Drug Metab Dispos. 2013 Aug;41(8):1488-93. doi: 10.1124/dmd.113.052316. Epub 2013 May 14. PMID 23674608
- [Background] Tomalik-Scharte D, Lutjohann D, Doroshyenko O, Frank D, Jetter A, Fuhr U. Plasma 4beta-hydroxycholesterol: an endogenous CYP3A metric? Clin Pharmacol Ther. 2009 Aug;86(2):147-53. doi: 10.1038/clpt.2009.72. Epub 2009 May 20. PMID 19458613
- [Background] Bergstrom H, Helde Frankling M, Klasson C, Lovgren Sandblom A, Diczfalusy U, Bjorkhem-Bergman L. CYP3A Activity in End-of-Life Cancer Patients Measured by 4beta-Hydroxycholesterol/cholesterol Ratio, in Men and Women. Cancers (Basel). 2021 Sep 18;13(18):4689. doi: 10.3390/cancers13184689. PMID 34572915
- [Background] Penzak SR, Rojas-Fernandez C. 4beta-Hydroxycholesterol as an Endogenous Biomarker for CYP3A Activity: Literature Review and Critical Evaluation. J Clin Pharmacol. 2019 May;59(5):611-624. doi: 10.1002/jcph.1391. Epub 2019 Feb 12. PMID 30748026
- [Background] Nylen H, Sergel S, Forsberg L, Lindemalm S, Bertilsson L, Wide K, Diczfalusy U. Cytochrome P450 3A activity in mothers and their neonates as determined by plasma 4beta-hydroxycholesterol. Eur J Clin Pharmacol. 2011 Jul;67(7):715-22. doi: 10.1007/s00228-010-0984-1. Epub 2011 Jan 19. PMID 21246351
- [Background] Naito T, Kubono N, Ishida T, Deguchi S, Sugihara M, Itoh H, Kanayama N, Kawakami J. CYP3A activity based on plasma 4beta-hydroxycholesterol during the early postpartum period has an effect on the plasma disposition of amlodipine. Drug Metab Pharmacokinet. 2015 Dec;30(6):419-24. doi: 10.1016/j.dmpk.2015.08.008. Epub 2015 Sep 3. PMID 26654672
- [Background] Kim AH, Kim B, Rhee SJ, Lee Y, Park JS, Lee SM, Kim SM, Lee S, Yu KS, Jang IJ, Cho JY. Assessment of induced CYP3A activity in pregnant women using 4beta-hydroxycholesterol: Cholesterol ratio as an appropriate metabolic marker. Drug Metab Pharmacokinet. 2018 Jun;33(3):173-178. doi: 10.1016/j.dmpk.2018.04.004. Epub 2018 Apr 25. PMID 29759884